CLINICAL TRIAL: NCT00592514
Title: Thyroid Dysfunction in Head and Neck Surgery Patients Treated With Intraoperative Oral Administration With Povidone-iodine 10% Solution
Brief Title: Thyroid Dysfunction in Head and Neck Surgery Patients
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 45976
Record Dates: First submitted 2007-12-27; First posted 2008-01-14 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Thyroid Dysfunction
Keywords: Patients undergoing head and neck surgery that involves the upper aerodigestive tract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Specific Aim I: Determine absorption of iodine after oropharyngeal application of povidone-iodine 10% solution when used in head and neck surgery involving the upper aero-digestive tract.

Specific Aim II: Measurement of iodine induced changes in thyroid function.

DETAILED DESCRIPTION:
Serial blood draws will be obtained from approximately 10 men and women age 18 and over who have been exposed to intraoperative oropharyngeal application with povidone-iodine 10%. Baseline serum and 24-hour urine iodine levels will be measured preoperatively. Serum iodine levels will be drawn at 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 1 week, and 1 month after exposure. A postoperative 24-hour urine iodine level will also be obtained. With the above measurements, the amount of iodine absorption as well as the time period of peak absorption and duration of elevated iodine levels will be elucidated.

Thyroid hormone metabolism is highly dependent on serum levels of iodine. Thyroid function will be assessed by measuring serum levels of free thyroxine, free triiodothyronine, and thyroid stimulating hormone also at 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 1 week, and 1 month after exposure. Measuring thyroid function is important since hypothyroidism has been known to have a major impact on postoperative wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing any head and neck surgery requiring entry into the upper aerodigestive tract and thus necessitating the oral administration of the antimicrobial agent povidone-iodine 10%.

Exclusion Criteria:

* Patients with history of hypothyroidism currently taking thyroid hormone medications (i.e. Synthroid, Levothyroxine, Thyroxine) and women who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Thyroid dysfunction in head and neck surgery patients | Baseline serum and 24-hour urine iodine levels will be measured preoperatively. Serum iodine levels will be drawn at 10 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours and 1 week after exposure.
  Specific Aim I: Determine absorption of iodine after oropharyngeal application of povidone-iodine 10% solution when used in head and neck surgery involving the upper aero-digestive tract.

SECONDARY OUTCOMES:
Thyroid dysfunction in head and neck surgery patients | Thyroid function will be assessed by measuring serum levels of free thyroxine, free triiodothyronine, and thyroid stimulating hormone also at 10 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours and 1 week after exposure.
  Specific Aim II: Measurement of iodine induced changes in thyroid function.

CONTACTS AND LOCATIONS:
Overall Officials: James Suen, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] 1. Betadine Solution [product label]. The Purdue Frederick Company. Stamford, CT. 2. Cannon, C. R. Hypothyroidism in head and neck cancer patients: experimental and clinical observations. Laryngoscope. 104(11 Pt 2 Suppl 66):1-21, 1994 Nov. 3. Ferguson, M., Geddes, D., Wray, D. The effect of a povidone-iodine mouthwash upon thyroid function and plaque accumulation. British Dental Journal. 144, 14, 1978. 4. Fradkin, J. E. and Wolff, J. Iodide-Induced Thyrotoxicosis. Medicine, 62, 1-20, 1983. 5. Guyétant, S., et al. Hyperthyroidism induced by amiodarone and hyperthyroidism induced by iodine. Histologic, immunohistochemical and ultrastructural aspects. Annales de Pathologie. 15(6):431-7, 1995.